CLINICAL TRIAL: NCT05851989
Title: Study on Prognosis of Acutely Ruptured Intracranial Aneurysms
Acronym: SPARTA
Status: Recruiting | Type: Observational
Sponsor: Haaglanden Medical Centre (Other)
Responsible Party: Principal Investigator, Wouter Moojen, Principal Investigator, Haaglanden Medical Centre
Other Study IDs: NL71261.058.19
Record Dates: First submitted 2023-02-22; First posted 2023-05-10 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage; Endovascular Procedures; Craniotomy; Patient Outcome Assessment; Treatment Outcome
Keywords: Aneurysmal subarachnoid hemorrhage; Clipping; Neurosurgery; Coiling; Endovascular treatment; Outcome; Modified Rankin Scale
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neurosurgical treatment: This cohort contains the patients with aneurysmal subarachnoid hemorrhage who received the neurosurgical clipping treatment.
- Endovascular treatment: This cohort contains the patients with neurysmal subarachnoid hemorrhage who received the endovascular coiling treatment. Other endovascular treatments which will be included as well are flow diverter procedures, Woven EndoBridge (WEB) devices and stent assisted coiling.

SUMMARY:
The SPARTA study is a prospective multicenter observational trial in the Netherlands with the aim of identifying the best clinical care in patients with aneurysmal subarachnoidal haemorrhage. Differences in outcome between surgical treatment and endovascular treatment will be explored.

Furthermore, cost effectiveness and radiological prognostic factors will be examined.

DETAILED DESCRIPTION:
Rationale:

Ruptured intracranial aneurysms resulting in subarachnoid haemorrhage can be treated by open surgical treatment or endovascular treatment. Despite multiple previous studies, biases and uncertainty around the best current treatment practice still exist. The resulting variation of care may result in a variable outcome. The protocol for a prospective multicentre observational study aimed at comparing the effectiveness of different treatment strategies in patients with ruptured aneurysms is presented.

Objective:

The primary aim of this study is to identify the effectiveness of clipping versus coiling on functional outcome in patients presenting with a subarachnoid haemorrhage due to a ruptured intracranial aneurysm 1 year after onset of symptoms. Secondary objectives include long term functional outcome, complications, cost-effectiveness and explorative analysis of the diagnostic and prognostic value of radiological imaging.

Study design:

This multi-centre study will have an observational prospective cohort design. Patient will have a follow-up of maximum 10 years.

Study population:

Patients with a subarachnoid haemorrhage will be included. Patients with evident other causes and patients without diagnosis of intracranial aneurysm after six months will be excluded.

Main study parameters/endpoints:

The primary endpoint is the score on the modified Rankin scale (mRs) and mortality at 1 year after the initial SAH. Secondary endpoints include the mRs, Modified Telephone Interview of Cognitive Status (TICS-M), 5-level EuroQol-5D (EQ-5D-5L) and derived Quality of Life Years, costs from patient diaries, and the Hospital Anxiety and Depression Scale (HADS), measured at 6 months, 1, 2, 5 and 10 years.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Patients will receive 'nonexperimental' regular care during their hospital stay. For this study, health questionnaires and functional outcome will be assessed at baseline, follow-up visits and before discharge. Temporary fatigue is the only possible side-effect of completion of the questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of subarachnoid haemorrhage on CT-scan or lumbar puncture (in the presence of a negative CT-scan)
* Intracranial aneurysm proven within 6 months to be the cause of subarachnoid haemorrhage
* Age 18 years or over at presentation.
* Written informed consent

Exclusion Criteria:

* Subarachnoid haemorrhage deemed most likely of 'perimesencephalic' origin after consideration of history, clinical examination and radiological findings (including angiographic imaging)
* Subarachnoid haemorrhage deemed most likely of post-traumatic origin after consideration of history, clinical examination and radiological findings (including angiographic imaging)
* Diagnosis of intracerebral arteriovenous malformations or dural arteriovenous fistula.
* No diagnosis of intracranial aneurysm at 6 months after onset of symptoms.
* Not mastering the Dutch language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that present primarily or after acute referral (in-patient to in-patient) to the participating centres, with a spontaneous subarachnoid haemorrhage will be screened for eligibility for this study by the treating physicians or local research nurses.
Sampling Method: Probability Sample
Enrollment: 880 (Estimated)
Dates: Start 2021-07-14 (Actual); Primary Completion 2025-07-14 (Estimated); Study Completion 2034-07-14 (Estimated)

PRIMARY OUTCOMES:
The score on the modified Rankin Scale at 1 year after onset of symptoms. | 1 year after onset of symptoms
  Scoring of functional outcome using the modified Rankin Scale. The scale has a minimum value of 0, meaning no symptoms, and a maximum value of 6, meaning dead. The modified Rankin Scale measures the degree of dependence. A higher score means a worse outcome.

SECONDARY OUTCOMES:
modified Rankin Scale at 6 months, 1, 2, 5 and 10 years after onset of symptoms, as measured by completion of case report forms by local treating teams | 6 months, 1, 2, 5 and 10 years after onset of symptoms
  Scoring of functional outcome using the modified Rankin Scale. The scale has a minimum value of 0, meaning no symptoms, and a maximum value of 6, meaning dead. The modified Rankin Scale measures the degree of dependence. A higher score means a worse outcome.
Modified Telephone Interview for Cognitive Status at 6 months, 1, 2, 5 and 10 years after onset as measured by completion of case report forms by local treating teams | 6 months, 1, 2, 5 and 10 years after onset of symptoms
  Scoring of cognitive outcome using the Modified Telephone Interview for Cognitive Status. This type of scoring contains multiple elements for detecting anamnestic mild cognitive impairment. The score ranges from 0 to 50, a higher score means a better outcome.
5-level EuroQol-5D questionnaire at 6 months, 1, 2, 5 and 10 years after onset of symptoms, as measured by completion of questionnaires by subjects | 6 months, 1, 2, 5 and 10 years after onset of symptoms
  Scoring of quality of life using the 5-level EuroQol-5D questionnaire. The questionnaire contains 5 scores in 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. A higher score means a worse outcome.
Health associated costs questionnaire | 3 months, 6 months, 1, 2, 5 and 10 years after onset of symptoms
  Estimation of societal costs by completion of a custom healthcare consumption and loss of productivity (paid and unpaid) questionnaire at 3 months, 6 months, 1 year, 2 years, 5 years and 10 years.

OTHER OUTCOMES:
Recanalization or recurrence of the treated aneurysm. | 6 months, 1, 2, 5 and 10 years after onset of symptoms
  Degree of occlusion in % of the aneurysm measured on imaging during follow-up using Computed Tomography, Diagnostic Angiography or Magnetic Resonance Imaging. A higher degree of occlusion means a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Wouter Moojen, MD, PhD, Principal Investigator — Haaglanden Medical Center
Locations (6):
- Netherlands (6):
  - Amsterdam UMC, Amsterdam
  - Maastricht UMC, Maastricht
  - Radboudumc, Nijmegen
  - Erasmus MC, Rotterdam
  - Haaglanden Medical Center, The Hague
  - Universitair Medisch Centrum Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hamming AL, van Dijck JTJM, Visser T, Baarse M, Verbaan D, Schenck H, Haeren RHL, Fakhry R, Dammers R, Aquarius R, Boogaarts JHD, Peul WC, Moojen WA. Study on prognosis of acutely ruptured intracranial aneurysms (SPARTA): a protocol for a multicentre prospective cohort study. BMC Neurol. 2024 Feb 17;24(1):68. doi: 10.1186/s12883-024-03567-6. PMID 38368355

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-04): https://cdn.clinicaltrials.gov/large-docs/89/NCT05851989/Prot_SAP_000.pdf